CLINICAL TRIAL: NCT01533181
Title: Randomized Phase II Study of Single Agent OSI-906, an Oral, Small Molecule, Tyrosine Kinase Inhibitor (TKI) of the Insulin Growth Factor-1 Receptor (IGF-1R) Versus Topotecan for the Treatment of Patients With Relapsed Small Cell Lung Cancer (SCLC)
Brief Title: Linsitinib or Topotecan Hydrochloride in Treating Patients With Relapsed Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NCI-2012-00245; NCI-2012-00245 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000724806; MCC-16628; MCC 16628 (Other: Moffitt Cancer Center); 8873 (Other: CTEP); N01CM00070 (NIH); N01CM00099 (NIH); N01CM00100 (NIH); P30CA076292 (NIH); NCT01387386 (obsolete NCT alias)
Record Dates: First submitted 2012-02-11; First posted 2012-02-15 (Estimated); Results first posted 2016-01-14 (Estimated); Last update posted 2016-01-14 (Estimated); Status verified 2015-08

CONDITIONS: Recurrent Small Cell Lung Carcinoma
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — 3-(8-amino-1-(2-phenylquinolin-7-yl)imidazo(1,5-a)pyrazin-3-yl)-1-methylcyclobutanol; Topotecan

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm I: OS-906 (linsitinib) (Experimental): OS-906 daily, continuously, every 3 weeks.
  Interventions: Other: Laboratory Biomarker Analysis; Drug: Linsitinib; Other: Pharmacological Study
- Arm II (topotecan hydrochloride) (Active Comparator): Patients receive topotecan hydrochloride IV over 30 minutes or PO QD on days 1-5. Patients may crossover to Arm I at the time of progressive disease.
  Interventions: Other: Laboratory Biomarker Analysis; Other: Pharmacological Study; Drug: Topotecan Hydrochloride

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Linsitinib — 150 mg given orally (PO) twice a day (BID)
  Other Names: IGF-1R inhibitor OSI-906; OSI-906; OSI-906AA
  Arms: Arm I: OS-906 (linsitinib)
Other: Pharmacological Study — Correlative studies
Drug: Topotecan Hydrochloride — 1.5 mg/m^2 intravenously (IV) or 2.3 mg/m^2 orally (PO)
  Other Names: Hycamptamine; Hycamtin; SKF S-104864-A; Topotecan HCl; topotecan hydrochloride (oral)
  Arms: Arm II (topotecan hydrochloride)

SUMMARY:
The purpose of this study is to evaluate how OSI-906 compares to Topotecan in trying to slow down the growth and/or progression of the tumors of participants with relapsed or recurrent Small Cell Lung Cancer.

This study also plans to find out what effects, good or bad (side effects), OSI-906 has on participants and or Small Cell Lung Cancer. The study will also investigate if some proteins measured in the blood or tumor and some imaging features obtained from computed tomography (CT) scans can help predict whether OSI-906 or topotecan will be effective against Small Cell Lung Cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To compare the progression-free survival (PFS) of single-agent OSI-906 (linsitinib) to that of single-agent topotecan (topotecan hydrochloride) in patients with relapsed small cell lung cancer (SCLC).

SECONDARY OBJECTIVES:

I. To evaluate the response rate (RR), disease-control rate (DCR) and overall survival (OS) of single-agent OSI-906 in patients with relapsed SCLC.

II. To describe the toxicity profile of single-agent OSI-906 in this population.

TERTIARY OBJECTIVES:

I. To evaluate potential predictive biomarkers of OSI-906 sensitivity. II. To determine whether the baseline insulin-like growth factor (IGF)-1, IGF-binding proteins (BPs), or angiogenic markers (vascular endothelial growth factor [VEGF] and interleukin [IL]-8) plasma levels or their pre- and post-treatment plasma level changes, significantly differ between progressor and non-progressor patients and correlate them with survival.

III. To assess whether the baseline protein kinase B (AKT) and/or mitogen-activated protein kinase 1 (ERK) phosphorylation or the extent of inhibition of AKT and/or ERK phosphorylation in peripheral blood mononuclear cells (PBMCs) significantly differs between progressors and non-progressors and to correlate them with survival.

IV. To determine whether the subcellular localization of IGF-1R, IGF-BPs, and/or the phosphorylation of IGF-1R throughout the cell by AQUA (automated quantitative immunofluorescence) significantly differs between progressors and non-progressors and correlate them with survival.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive linsitinib orally (PO) twice daily (BID) on days 1-21.

ARM II: Patients receive topotecan hydrochloride intravenously (IV) over 30 minutes or PO once daily (QD) on days 1-5. Patients may crossover to Arm I at the time of progressive disease.

In both arms, courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 4 weeks and then every 6 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed SCLC
* Patients must have measurable disease; at least one lesion that can be accurately measured is required
* Patients must have progression of disease after receiving ONLY 1 previous platinum-containing regimen; prior treatment with biological response modifiers or targeted agents will NOT count towards this requirement; previous topotecan or any type of pharmacologic IGF-1R inhibition are NOT allowed
* Life expectancy of greater than 6 weeks
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) =< 2; (Karnofsky >= 60%)
* Leukocytes (white blood cell [WBC]) >= 3,000/mcL OR
* Absolute neutrophil count (ANC) >= 1,500/mcL
* Platelets >= 100,000/mcL
* Total bilirubin within normal institutional limits (NIL)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.0 times institutional upper limit of normal (ULN) without demonstrable liver metastases OR < 5.0 times ULN with liver metastases present
* Serum creatinine within NIL OR measured/calculated creatinine clearance (CrCl) >= 60 mL/min/1.73 m^2 for patients with creatinine levels above NIL
* Fasting blood glucose < 160 mg/dL at baseline
* Patients on oral antihyperglycemic therapies may be enrolled provided they have been taking a stable dose of these medications for >= 2 weeks at the time of randomization
* Prior radiation is permitted IF the site(s) of measurable disease has progressed since prior irradiation and radiation is completed at least 2 weeks before initiation of drug treatment (stereotactic radiotherapy excluded)
* Patients with central nervous system (CNS) metastases are ELIGIBLE, provided that prior to drug treatment, the metastases have been treated, remain clinically or radiographically stable and the patient has no significant neurologic symptoms
* Patients must NOT have prior malignancy EXCEPT for the following: adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, adequately treated stage I or II cancer from which the patient is currently in complete remission, or any other cancer from which the patient has been disease-free for >= 3 years
* Women of child-bearing potential (WOCBP) and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately; WOCBP must provide a negative pregnancy test (serum or urine) within 14 days prior to registration
* Available archival tumor tissue is NOT mandatory for enrollment (will be requested)
* Patients must have the ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients who have had chemotherapy within 3 weeks (6 weeks for nitrosoureas or mitomycin C) or radiotherapy within 2 weeks prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier
* Patients who are receiving any other investigational agents
* Patients with CNS metastases are NOT EXCLUDED, provided that prior to drug treatment, the metastases have been treated, remain radiographically stable and the patient has no significant neurologic symptoms
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to OSI-906 or other agents used in the study (topotecan)
* While cytochrome P450, family 1, subfamily A, polypeptide 2 (CYP1A2) inhibitors/inducers are not specifically excluded, investigators should be aware that the metabolism and consequently overall pharmacokinetics (PKs) of OSI-906 (OSI-906 exposure) could be altered by concomitant use of these drugs (inhibitors, inducers and/or other substrates of CYP1A2); exception: potent CYP1A2 inhibitors ciprofloxacin and fluvoxamine are prohibited; while cytochrome P450, family 2, subfamily C, polypeptide 9 (CYP2C9) substrates are not specifically excluded, investigators should be aware that levels of drugs metabolized by CYP2C9 may be increased by the concomitant administration of OSI-906; caution should be used when administering CYP2C9 substrates to study patients
* The concomitant use of p-glycoprotein inhibitors with topotecan capsules is not allowed
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, significant cardiac disease (i.e., symptomatic congestive heart failure, unstable angina pectoris, symptomatic or life-threatening cardiac arrhythmia), or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant or breast-feeding women are excluded from this study
* Human immunodeficiency virus (HIV)-positive patients on combination antiretroviral therapy are ineligible
* Patients in the following scenarios are excluded:

  * Corrected QT (QTc) interval > 450 msec at baseline
  * Concomitant drugs that prolong the QTc interval
  * Use of drugs that have a known risk of causing Torsades de Pointes (TdP) within 14 days prior to randomization
  * Fasting blood glucose >= 160 mg/dL at baseline; these patients can initiate allowed oral antihyperglycemic therapies and be retested or rescreened 2 weeks later to meet baseline fasting blood glucose criteria
  * Concomitant use of insulin or insulinotropic medications
* Patients with cirrhosis of the liver are excluded from this study
* Archival tumor tissue is NOT mandatory for enrollment, but will be requested

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2012-02; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alberto Chiappori, Principal Investigator — Moffitt Cancer Center
Locations (11):
- United States (10):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Moffitt Cancer Center, Tampa, Florida
  - Emory University/Winship Cancer Institute, Atlanta, Georgia
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins Hospital, Baltimore, Maryland
  - Billings Clinic Cancer Center, Billings, Montana
  - Case Western Reserve University, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
- Johns Hopkins Singapore, Singapore, Singapore

REFERENCES:
- [Derived] Chiappori AA, Otterson GA, Dowlati A, Traynor AM, Horn L, Owonikoko TK, Ross HJ, Hann CL, Abu Hejleh T, Nieva J, Zhao X, Schell M, Sullivan DM. A Randomized Phase II Study of Linsitinib (OSI-906) Versus Topotecan in Patients With Relapsed Small-Cell Lung Cancer. Oncologist. 2016 Oct;21(10):1163-1164. doi: 10.1634/theoncologist.2016-0220. Epub 2016 Sep 30. PMID 27694157

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at Moffitt Cancer Center and nine other institutions in the United States from July 3, 2012 through November 1, 2013.
Groups:
- Arm A: Topotecan: Participants receive topotecan hydrochloride IV over 30 minutes or orally (PO) daily (QD) on days 1-5. Patients may crossover to Arm B at the time of progressive disease.
- Arm B: OS-906: OS-906 (linsitinib) daily, continuously, every 3 weeks.
Period: Overall Study
Arm/Group | Arm A: Topotecan | Arm B: OS-906
Started | 15 | 29
Completed | 14 | 28
Not Completed | 1 | 1
Not completed — Disease progression pre-active treatment | 0 | 1
Not completed — Patient withdrawal pre-active treatment | 1 | 0

BASELINE CHARACTERISTICS:
Population: All participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A: Topotecan | Arm B: OS-906 | Total
Number analyzed (Participants) | 15 | 29 | 44
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 9 | 17 | 26
  >=65 years | 6 | 12 | 18
Age, Continuous [Median (Full Range); unit: years] | 64 [34 to 86] | 62 [37 to 79] | 64 [34 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 17 | 25
  Male | 7 | 12 | 19
Region of Enrollment [Number; unit: participants]
  United States | 15 | 29 | 44

OUTCOME MEASURES:

1. Primary Outcome: Median Progression Free Survival (PFS)
Description: PFS: Time from randomization to time of disease progression or death. PFS summarized with the Kaplan-Meier (K-M) method by two arms (experimental versus control). Confidence intervals for the median PFS and PFS rates at different time points to be constructed when appropriate.
Time Frame: Up to 6 months
Population: All participants who received treatment
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A: Topotecan | Arm B: OS-906
Number analyzed (Participants) | 14 | 28
months | 3 [1.5 to 3.6] | 1.2 [1.1 to 1.4]
Statistical Analysis 1: Comparison: Arm A: Topotecan vs Arm B: OS-906; Test type: Superiority or Other; p = 0.0001, Kaplan-Meier; Hazard Ratio (HR) = 3.9, 95% CI 2-sided [1.9 to 8.1]

2. Secondary Outcome: Disease Control Rate (DCR)
Description: DCR: Complete Response (CR) + Partial Response (PR) + Stable Disease (SD) + Progressive Disease (PD). DCR summarized using both point estimates and exact confidence intervals based on the binomial distribution by arm.
Time Frame: Up to 2 years
Population: All evaluable participants at time of analysis
Measure: Number; unit: participants
Arm/Group | Arm A: Topotecan | Arm B: OS-906
Number analyzed (Participants) | 12 | 25
participants
  Complete Response | 0 | 0
  Partial Response | 2 | 0
  Stable Disease | 4 | 1
  Progressive Disease | 6 | 24
  Disease Control Rate | 6 | 1

3. Secondary Outcome: Incidence of Serious Adverse Events (SAEs) Possibly/Probably Definitely Related to Study Drugs
Description: Participants with Grade 3 and 4 toxicities, possibly/probably/definitely related to study drugs. Number of Participants is per Event Category. Assessed by National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0.
Time Frame: 1 year, 6 months
Population: All participants who received treatment
Measure: Number; unit: participants
Arm/Group | Arm A: Topotecan | Arm B: OS-906
Number analyzed (Participants) | 14 | 28
participants
  Anemia | 1 | 1
  Blood and lymphatic system disorders - Other | 2 | 0
  Thrombotic thrombocytopenic purpura | 1 | 0
  Diarrhea | 1 | 0
  Esophagitis | 1 | 0
  Pancreatitis | 1 | 0
  Fatigue | 1 | 3
  Alanine aminotransferase increased | 0 | 2
  Investigations - Other | 1 | 0
  Lymphocyte count decreased | 2 | 3
  Neutrophil count decreased | 4 | 0
  Platelet count decreased | 4 | 2
  White blood cell decreased | 4 | 0
  Anorexia | 0 | 1
  Dehydration | 2 | 0
  Hyperglycemia | 0 | 1
  Hypokalemia | 1 | 0
  Hyponatremia | 0 | 1
  Headache | 0 | 1
  Hypoxia | 0 | 1
  Thromboembolic event | 1 | 0

4. Secondary Outcome: Overall Survival (OS)
Description: OS: Time from study enrollment to death from any cause. OS summarized similarly to PFS utilizing the K-M method.
Time Frame: Up to 2 years
Population: All participants who received treatment
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A: Topotecan | Arm B: OS-906
Number analyzed (Participants) | 14 | 28
months | 5.3 [2.2 to 7.6] | 3.4 [1.8 to 5.6]
Statistical Analysis 1: Comparison: Arm A: Topotecan vs Arm B: OS-906; Test type: Superiority or Other; p = 0.71, Kaplan-Meier; Hazard Ratio (HR) = 1.1, 95% CI 2-sided [0.6 to 2.2]

5. Other Pre Specified Outcome: Changes in Biomarker Expression
Description: To be assessed by the Wilcoxon rank sum test.
Time Frame: Baseline to up to day 1 of course 3
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 1 year, 6 months
Description: Adverse Events are reported for all participants who received treatment, regardless of causality.
  Grades 3, 4 and 5 are noted on the appropriate reported SAEs.
  Note: Causality for SAEs is addressed in the Secondary Outcome Measure area.
Groups:
- Arm A: Topotocan: Participants receive topotecan hydrochloride IV over 30 minutes or orally (PO) daily (QD) on days 1-5. Patients may crossover to Arm B at the time of progressive disease.
Arm/Group | Arm A: Topotocan | Arm B: OS-906
Serious Adverse Events (participants affected / at risk) | 7/14 | 18/28
Other Adverse Events (participants affected / at risk) | 12/14 | 28/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: Topotocan (N=14) | Arm B: OS-906 (N=28)
Anemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) — Arm A: 1 Grade 3 event
Blood and lymphatic system disorders - Other, Pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) — Grade 4
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) — Grade 3
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) — Grade 3
Esophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0) — Grade 3
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) — Grade 3
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Death NOS (General disorders) | 7 (7) | 12 (12) — No Death SAE was due to treatment. All due to disease progression. Grade 5
Fever (General disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1) — Grade 3
Pain (General disorders) | 0 (0) | 1 (1) — Grade 3
Enterocolitis infectious (Infections and infestations) | 1 (1) | 0 (0) — Grade 3
Infections and infestations - Other, Possible pneumonia per x-ray (Infections and infestations) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 3 (4) — 3 Grade 3, 1 Grade 5
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) — Grade 3
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) — Grade 3
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Blood bilirubin increase (Investigations) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 0 (0) | 1 (1) — Grade 4
Neutrophil count decreased (Investigations) | 1 (1) | 0 (0) — Grade 4
Platelet count decreased (Investigations) | 0 (0) | 1 (1) — Grade 3
White blood cell decreased (Investigations) | 2 (2) | 0 (0) — Grade 4
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 2 (2) — Arm A: Grade 3
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) — Grade 3
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) — Grade 4
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — Grade 3
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — Grade 3
Neoplasms benign, malignant and unspecified - Other, Progressive disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 3 (3) — Grade 4
Neoplasms benign, malignant and unspecified - Other, Death (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 6 (6) — No Death SAE was due to treatment. All due to disease progression. Grade 5
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) — Grade 3
Headache (Nervous system disorders) | 0 (0) | 1 (1) — Grade 3
Intracranial hemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 1 (1)
Confusion (Psychiatric disorders) | 1 (1) | 1 (1) — Grade 3
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (6) — 5 events were Grade 3
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) — Grade 3
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Grade 5
Respiratory, thoracic and mediastinal disorders - Other, COPD (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Grade 3
Hypotension (Vascular disorders) | 1 (1) | 0 (0) — Grade 3
Superior vena cava syndrome - Death (Vascular disorders) | 0 (0) | 1 (1) — No Death SAE was due to treatment. All due to disease progression. Grade 5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: Topotocan (N=14) | Arm B: OS-906 (N=28)
Fatigue (General disorders) | 8 (11) | 16 (18)
Pain (General disorders) | 3 (3) | 6 (8)
Chills (General disorders) | 1 (1) | 2 (2)
Fever (General disorders) | 2 (2) | 0 (0)
General Disorders - Other (General disorders) | 1 (1) | 2 (2)
Flu like symptoms (General disorders) | 0 (0) | 2 (2)
Malaise (General disorders) | 1 (1) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 2 (2)
Edema face (General disorders) | 0 (0) | 1 (1)
Edema limbs (General disorders) | 0 (0) | 1 (1)
Edema trunk (General disorders) | 1 (1) | 0 (0)
Facial pain (General disorders) | 0 (0) | 1 (1)
Gait disturbance (General disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 6 (7) | 13 (15)
Vomiting (Gastrointestinal disorders) | 6 (8) | 8 (10)
Constipation (Gastrointestinal disorders) | 5 (5) | 8 (9)
Diarrhea (Gastrointestinal disorders) | 3 (4) | 6 (8)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 0 (0) | 4 (4)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 3 (3)
Mucositis oral (Gastrointestinal disorders) | 2 (2) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 2 (2)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 1 (1)
Bloating (Gastrointestinal disorders) | 0 (0) | 1 (1)
Fecal incontinence (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oral hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oral pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Stomach pain (Gastrointestinal disorders) | 1 (2) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 7 (7) | 12 (13)
Hyponatremia (Metabolism and nutrition disorders) | 2 (2) | 11 (19)
Hyperglycemia (Metabolism and nutrition disorders) | 3 (3) | 8 (10)
Hypoalbuminemia (Metabolism and nutrition disorders) | 4 (4) | 8 (14)
Dehydration (Metabolism and nutrition disorders) | 4 (6) | 4 (4)
Hypokalemia (Metabolism and nutrition disorders) | 2 (2) | 6 (9)
Hypocalcemia (Metabolism and nutrition disorders) | 2 (2) | 5 (5)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1) | 2 (4)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Metabolism and nutrition disorders - Other (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Alkalosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 1 (3)
Hypernatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 8 (10)
White blood cell decreased (Investigations) | 7 (14) | 2 (5)
Alanine aminotransferase increased (Investigations) | 1 (1) | 7 (9)
Lymphocyte count decreased (Investigations) | 5 (15) | 5 (15)
Platelet count decreased (Investigations) | 4 (9) | 4 (7)
Blood bilirubin increased (Investigations) | 1 (1) | 6 (6)
Weight loss (Investigations) | 0 (0) | 6 (6)
Alkaline phosphatase increased (Investigations) | 0 (0) | 5 (6)
Neutrophil count decreased (Investigations) | 5 (8) | 0 (0)
Creatinine increased (Investigations) | 0 (0) | 4 (7)
Electrocardiogram QT corrected interval prolonged (Investigations) | 1 (1) | 1 (1)
INR increased (Investigations) | 1 (1) | 1 (1)
Investigations - Other (Investigations) | 2 (3) | 1 (1)
Cardiac troponin I increased (Investigations) | 1 (1) | 0 (0)
CD4 lymphocytes decreased (Investigations) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 8 (8)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 6 (6)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (4)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 11 (25) | 7 (12)
Blood and lymphatic system disorders - Other (Blood and lymphatic system disorders) | 2 (2) | 2 (2)
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 2 (4) | 3 (3)
Headache (Nervous system disorders) | 3 (5) | 2 (5)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 3 (3)
Lethargy (Nervous system disorders) | 0 (0) | 1 (1)
Amnesia (Nervous system disorders) | 1 (1) | 0 (0)
Dysarthria (Nervous system disorders) | 0 (0) | 1 (3)
Nervous system disorders - Other (Nervous system disorders) | 1 (1) | 0 (0)
Paresthesia (Nervous system disorders) | 0 (0) | 1 (1)
Phantom pain (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (7)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (4)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (4)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 4 (4)
Hypertension (Vascular disorders) | 2 (3) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (4) | 1 (1)
Vascular disorders - Other (Vascular disorders) | 2 (2) | 0 (0)
Flushing (Vascular disorders) | 1 (1) | 2 (2)
Hot flashes (Vascular disorders) | 0 (0) | 1 (1)
Superior vena cava syndrome (Vascular disorders) | 0 (0) | 1 (2)
Neoplasms benign, malignant and unspecified - Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 8 (8)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Hypohidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Infections and infestations - Other (Infections and infestations) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (2)
Vaginal infection (Infections and infestations) | 0 (0) | 1 (1)
Confusion (Psychiatric disorders) | 2 (2) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 2 (2)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 1 (2)
Tinnitus (Ear and labyrinth disorders) | 1 (2) | 0 (0)
Eyelid function disorder (Eye disorders) | 0 (0) | 1 (1)
Watering eyes (Eye disorders) | 0 (0) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Allergic reaction (Immune system disorders) | 0 (0) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less